CLINICAL TRIAL: NCT02325271
Title: Intra-individual Variability and Circadian Rhythm of Systemic Vascular Endothelial Growth Factor (VEGF) Levels and Interaction With Biomarkers of Inflammation in Subjects With Normal Glucose Tolerance (NGT) and Patients With Type 2 Diabetes Without Diabetic Macular Edema (DME)
Brief Title: Intra-individual Variability and Circadian Rhythm of VEGF Levels and Interaction With Biomarkers
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: VEGF Bio
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Subjects with normal glucose tolerance
  Interventions: Other: Frequent blood and urine sampling and blood pressure measurement
- Diabetes group: Patients with type 2 diabetes
  Interventions: Other: Frequent blood and urine sampling and blood pressure measurement

INTERVENTIONS:
Other: Frequent blood and urine sampling and blood pressure measurement — Blood and urine sampling for the determination of VEGF and biomarkers

SUMMARY:
The study evaluates the intra-individual variability of VEGF levels over a period of 6 months as well as the circadian variation of VEGF levels, both under standardized conditions in patients with type 2 diabetes without DME and matched subjects with normal glucose tolerance (NGT). Secondary objectives of the study are to evaluate the relationship of individual VEGF-levels to biomarkers of inflammation, HbA1c and major cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age equal to or between 50 and 80 years
* Subjects with normal glucose tolerance confirmed by glucose tolerance test (control group) or patients with type 2 diabetes: diabetes duration 5-25 years; HbA1c equal to or between 6.5 and 9% (diabetes group)
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* DME
* hsCRP > 10 mg/dl
* Acute infections
* Acute or chronic inflammatory diseases
* Immune diseases
* Treatment with immune suppressive drugs
* Treatment with glucocorticoids
* Myocardial infarction and stroke within 1 year before inclusion
* Hemorrhage within the previous 5 years
* Surgeries within the previous 3 months
* Oncological diseases
* Women who are pregnant or breast-feeding

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample of healthy volunteers, type 2 diabetes patients of the study center
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
VEGF-A | Baseline, month 1, 2, 3, 4, 5 and 6
  Plasma levels determined in the morning under fasted conditions
VEGF-B | Baseline, month 1, 2, 3, 4, 5 and 6
  Plasma levels determined in the morning under fasted conditions
VEGF-C | Baseline, month 1, 2, 3, 4, 5 and 6
  Plasma levels determined in the morning under fasted conditions
Placental growth factor | Baseline, month 1, 2, 3, 4, 5 and 6
  Plasma levels determined in the morning under fasted conditions
VEGF-A | Hourly over 12 hours
  Plasma levels determined over the day
VEGF-B | Hourly over 12 hours
  Plasma levels determined over the day
VEGF-C | Hourly over 12 hours
  Plasma levels determined over the day
Placental growth factor | Hourly over 12 hours
  Plasma levels determined over the day

SECONDARY OUTCOMES:
Glycated hemoglobin (HbA1c) | Baseline, month 1, 2, 3, 4, 5 and 6
  Plasma levels determined in the morning under fasted conditions
High-sensitivity C-reactive protein (hCRP) | Baseline, month 1, 2, 3, 4, 5 and 6
  Serum levels determined in the morning under fasted conditions
Matrix metallopeptidase 9 (MMP-9) | Baseline, month 1, 2, 3, 4, 5 and 6
  Plasma levels determined in the morning under fasted conditions
MMP-9 | Hourly over 12 hours
  Plasma levels determined over the day
Adiponectin | Baseline, month 1, 2, 3, 4, 5 and 6
  Serum levels determined in the morning under fasted condition
Adiponectin | Hourly over 12 hours
  Serum levels determined over the day
Cystatin C | Baseline, month 1, 2, 3, 4, 5 and 6
  Serum levels determined in the morning under fasted condition
Cystatin C | Hourly over 12 hours
  Serum levels determined over the day
Albumin | Baseline, month 1, 2, 3, 4, 5 and 6
  Urine levels determined in the morning under fasted condition
Creatinine | Baseline, month 1, 2, 3, 4, 5 and 6
  Urine levels determined in the morning under fasted condition
Creatinine | Baseline, month 1, 2, 3, 4, 5 and 6
  Serum levels determined in the morning under fasted condition
Blood pressure | Baseline, month 1, 2, 3, 4, 5 and 6, once over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Markolf Hanefeld, Prof. Dr., Principal Investigator — Study center Prof. Hanefeld, GWT-TUD GmbH
Locations (1):
- GWT-TUD GmbH / Studienzentrum Hanefeld, Dresden, Germany

REFERENCES:
- [Derived] Hanefeld M, Engelmann K, Appelt D, Sandner D, Weigmann I, Ganz X, Pistrosch F, Kohler C, Gasparic A, Birkenfeld AL. Intra-individual variability and circadian rhythm of vascular endothelial growth factors in subjects with normal glucose tolerance and type 2 diabetes. PLoS One. 2017 Oct 9;12(10):e0184234. doi: 10.1371/journal.pone.0184234. eCollection 2017. PMID 28991900